CLINICAL TRIAL: NCT05771961
Title: Impact of Rotational Atherectomy on Coronary Microvascular Function in Patients With Stable Angina and Calcified Coronary Artery Disease
Brief Title: Impact of Rotational Atherectomy on Coronary Microcirculation
Acronym: MICRO-ROTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Klaipėda University (Other); Kreiskrankenhaus Rotenburg an der fluda (Unknown); Alkafeel Super Speciality Hospital (Unknown)
Responsible Party: Principal Investigator, Ali Aldujeli, Cardiovascular disease consultant, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUHSKC-179
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Stable Angina; Coronary Artery Disease
Keywords: Rotational atherectomy; Conventional stenting; CMD; Microcirculation; Index of microcirculatory resistance; IMRangio
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to receive either the rotational atherectomy or conventional stenting alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational Atherectomy (Active Comparator): Patients who are scheduled to have rotational atherectomy will be labeled in this group; patients in this group will have invasive and non-invasive microvascular testing before and after the rotational atherectomy procedure.
  Interventions: Diagnostic Test: coronary pressure/temperature sensor-tipped guidewire; Diagnostic Test: Angiography-derived index of microcirculatory resistance (IMRangio)
- Conventional Stenting (Active Comparator): Patients who are scheduled to have conventional stenting will be labeled in this group; patients in this group will have invasive and non-invasive microvascular testing before and after the conventional stenting procedure.
  Interventions: Diagnostic Test: coronary pressure/temperature sensor-tipped guidewire; Diagnostic Test: Angiography-derived index of microcirculatory resistance (IMRangio)

INTERVENTIONS:
Diagnostic Test: coronary pressure/temperature sensor-tipped guidewire — In brief, a 6-F angioplasty guiding catheter without side-holes will be used first used to engage the left main coronary artery. A pressure-temperature sensor guidewire ( PressureWire™ X Guidewire) will be used for physiology measurements including IMR measurements.
  Pressure measurement from the wire will be first equalized with that of the guiding catheter. Then the pressure sensor will be positioned two-thirds of the way down the LAD artery. Intracoronary nitroglycerin will be administered (100 to 200 μg). Hyperemia will be induced with adenosine intracoronary injections.
Diagnostic Test: Angiography-derived index of microcirculatory resistance (IMRangio) — Angiography-derived index of microcirculatory resistance (IMRangio) will be calculated by an anticipated software

SUMMARY:
The purpose of this observational study is to compare the impact of rotational atherectomy to conventional stenting and to investigate how it may affect coronary microcirculation in patients with calcified coronary artery lesions and stable CAD.

The study's objectives are to:

* investigate the impact of rotational atherectomy on the prevalence of post-percutaneuos coronary intervention coronay microvascular dysfunction;
* investigate the impact of conventional stenting on the prevalence of post-percutaneuos coronary intervention coronay microvascular dysfunction; and
* compare the impact of both percutaneuos coronary interventions on coronary microvascular dysfunction.

Patients with calcified lesions will be enrolled prospectively and will have serial invasive and non-invasive microvascular testing prior to and after rotational atherectomy or conventional stenting.

DETAILED DESCRIPTION:
Rotational atherectomy (RA) is a medical procedure used to treat patients with severe atherosclerosis, a condition that causes plaque buildup within the artery walls, resulting in narrowing of the blood vessels and decreased blood flow to the heart. RA is a technique that involves breaking up and removing plaque from the artery with a small, high-speed rotating burr.

However, RA is not without risks. One of the major risks associated with RA is the potential damage to the artery wall and surrounding tissue. This can lead to complications such as bleeding, blood clots, or injury to the heart or other organs. Additionally, the high-speed rotation of the burr can generate heat, which may damage the artery wall or cause the release of harmful particles into the bloodstream.

Another hypothesized risk of RA is its impact on microcirculation, which refers to the smallest blood vessels in the body. RA can cause disruption to these vessels, leading to a decrease in blood flow and potentially causing damage to tissues and organs that depend on them.

The purpose of this study is to look into the effect of rotational atherectomy on coronary microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with stable coronary artery calcified lesion requiring Percutaneous coronary intervention

Exclusion Criteria:

* patients with a history of old myocardial infarction or history of coronary artery bypass grafting (CABG) or Percutaneous coronary intervention PCI
* Patients with signs of chronic infection, prolong usage of corticosteroids or compromised immune system
* patients had contraindication of adenosine triphosphate (ATP);
* had a history of liver or renal function dysfunction
* Patients with dementia
* Patients being referred to CABG
* unable to provide informed consent;
* had pregnancy or life span < 1 year.
* Presence of sever structural valvular heart disease
* Presence of significant left main disease
* Unability to measure the index of microcirculatory resistance due to (death or retraction from the study ...etc)
* Inability to perform successful PCI

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of coronary microvascular dysfunction | 1 day
  Microcirculatory dysfunction will be defined as having an IMR value ≥ 25 U and a CFR value < 2.5 U or angio IMR ≥ 25 U

SECONDARY OUTCOMES:
Rate of Major adverse cardiovascular events | 1 year
  composite of nonfatal stroke, nonfatal myocardial infarction, heart failure, target vessel revascularization and cardiovascular death.
The incidence of coronary microvascular dysfunction | 1 year
  Microcirculatory dysfunction will be defined as having an IMR value ≥ 25 U and a CFR value < 2.5 U or angio IMR ≥ 25 U
Seattle Angina Questionnaire score | 1 year
  Evaluates the severity of angina symptoms, physical limitations, and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aldujeli, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided